CLINICAL TRIAL: NCT03763266
Title: Low Residue Diet 3 Days Versus 1 Day as Preparation for Colonoscopy: a Randomized Controlled Trial
Brief Title: Low Residue Diet During 3 Days vs 1 Day Prior Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Salvador Machlab, Principal Investigator, Parc Taulí Hospital Universitari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2017308
Record Dates: First submitted 2018-11-10; First posted 2018-12-04 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Colonoscopy; Colon Adenoma; Colorectal Neoplasms; Inflammatory Bowel Diseases; Colon Disease
Keywords: bowel preparation; low residue diet; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Colonic Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 day low residue diet (Experimental): Patients are instructed to complete a low residue diet exclusively one day prior the colonoscopy.
  Interventions: Other: 1 day low residue diet
- 3 days low residue diet (Active Comparator): Patients are instructed to complete a low residue diet three days prior the colonoscopy.
  Interventions: Other: 3 day low residue diet

INTERVENTIONS:
Other: 1 day low residue diet — Patients are interviewed and instructed by a nurse prior the colonoscopy. They receive oral and written dietary information. In case of morbidity associated with bad preparation they are given bisacodyl the night before the colonoscopy.
  Other Names: low fiber diet
  Arms: 1 day low residue diet
Other: 3 day low residue diet — Patients are interviewed and instructed by a nurse prior the colonoscopy. They receive oral and written dietary information. In case of morbidity associated with bad preparation they are given bisacodyl the night before the colonoscopy.
  Other Names: low fiber diet
  Arms: 3 days low residue diet

SUMMARY:
Colonoscopy is the gold-standard for the evaluation of the colorectal mucosa. Colonoscopy quality indicators are the adenoma detection rate, the rate of cecal intubation and the bowel preparation.

The role of diet in preparing for colonoscopy is not fully established. Currently there is not enough evidence available to choice between 3 days of low residue diet versus 1 day.

The research hypothesis is that the low residue diet offers a non-inferior bowel preparation and an improved tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the colorectal cancer screening program that give consent

Exclusion Criteria:

* Contraindication for colonoscopy

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Bowel preparation | During the colonoscopy
  Measured with the Boston Bowel Preparation Scale from 0 until 9. 9 represents an excellent preparation.

SECONDARY OUTCOMES:
Diet tolerance | It is reported before entering the endoscopy room. Regarding the 3 or 1 days on low fiber diet depending on which study group is the participant.
  Using Likert scale. From 1 to 5, lower is better tolerance.
Preparation tolerance | It is reported before entering the endoscopy room. Regarding the 3 or 1 day on bowel preparation depending on which study group is the participant.
  Using Likert scale. From 1 to 5, lower is better tolerance.
Adenoma detection rate | up to 2 weeks after colonoscopy depending on pathology department workload.
  Proportion of colonoscopies with detection of colorectal cancer or adenoma excluding distal hyperplastic
Endoscopic diagnosis | It is assessed during the colonoscopy and will be reported the same day.
  Final endoscopic diagnosis. For example; normal, diverticulosis, polyps, colorectal cancer, etc.
Cecum intubation rate | It will be calculated through study completion, approximately 1 year, for all the study period using all participants having the colonoscopy done
  Cecum intubation will be assessed during each colonoscopy if the endoscope reaches the cecum.
Intubation time | it is assessed from the start of the colonoscopy until cecum is reached (1 day)
  time lapse from the start of the exploration until cecum is reached.
Withdrawal time | it is assessed from at the beginning of the withdrawal of the colonoscope until the colonoscopy is finished. (procedure)
  Time lapse between cecum withdrawal the end of the exploration.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Martínez, PhD, Study Director — Corporació Sanitaria Parc Taulí; Salvador Machlab, MD, Principal Investigator — Corporació Sanitaria Parc Taulí; Rafel Campo, PhD, Study Director — Corporació Sanitaria Parc Taulí
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain